CLINICAL TRIAL: NCT03271008
Title: Comparison of Necessary Time for Successful Intubation With the Vividtrac™ and KingVision™ Videolaryngoscopes and Macintosh Blade Direct Laryngoscopy in Clinical Practice
Brief Title: Comparison of the Vividtrac™ and Other Videolaryngoscopes in Clinical Practice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Gábor László Woth, clinical resident, PhD, University of Pecs
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 6328
Record Dates: First submitted 2017-05-11; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Intubation;Difficult

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Following informed consent participants are randomised into one of the device groups and general anaesthesia is induced. Primary intubation attempt is carried out with the randomised device. We do not disclose the result of randomisation with our participants prior to anaesthesia induction. Participants are already in surgical anaesthesia with muscle relaxation during the intubation attempt. As providers are the users of the intubation device masking is not possible in this regard. During outcome assessment we plan not to disclose which device was used for a certain group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Macintosh laryngoscopy (Active Comparator): In this group intubation attempt is carried out with a standard Macintosh (size 3 or 4) direct laryngoscopy blade.
  Interventions: Device: Direct laryngoscopy
- KingVision videolaryngoscope (Active Comparator): In this group intubation attempt is carried out with KingVision videolaryngoscope with a channeled, disposable single-use blade.
  Interventions: Device: KingVision videolaryngoscope
- VividTrac videolaryngoscope (Active Comparator): In this group intubation attempt is carried out with VividTrac Adult model using a smartphone or laptop running the VividVision proprietary software.
  Interventions: Device: Vividtrac videolaryngoscope

INTERVENTIONS:
Device: Direct laryngoscopy — During the induction of general anaesthesia, the first attempt to achieve a secured airway is carried out using a size 4 (or size 3 if necessary) Macintosh blade direct laryngoscope.
  Arms: Macintosh laryngoscopy
Device: Vividtrac videolaryngoscope — During the induction of general anaesthesia, the first attempt to achieve a secured airway is carried out using a Vividtrac videolaryngoscope connected to a tablet or smartphone.
  Arms: VividTrac videolaryngoscope
Device: KingVision videolaryngoscope — During the induction of general anaesthesia, the first attempt to achieve a secured airway is carried out using a KingVision videolaryngoscope.
  Arms: KingVision videolaryngoscope

SUMMARY:
Comparison of various videolaryngoscope devices (Vividtrac™ and KingVision™) and direct laryngoscopy with Macintosh blade regarding laryngoscopy time, intubation time, intubation success rate, percentage of visible glottic opening (POGO score) in elective and acute clinical anaesthesiology practice.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* over 18 years of age
* elective intervention
* no anticipated difficult airway or intubation
* preoperative anaesthesia risk assessment by American Society of Anaesthesiologists (ASA) physical status classification: ASA grade I-II

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Intubation time | Measured once during the intubation attempt. Up to 120 seconds following the start of intubation attempt.
  Time necessary to secure airway during the induction of general anesthesia. Intubation time is measured from the point the airway device crosses the interdental line until the completion of intubation with insufflated cuffed endotracheal tube (secured airway).

SECONDARY OUTCOMES:
Laryngoscopy time | Registered once during the intubation attempt. Up to 120 seconds following the start of intubation attempt.
  Time necessary to achieve best visualisation of the glottic opening.
Percentage of glottic opening (POGO) score | Registered once during the intubation attempt. Up to 120 seconds following the start of intubation attempt.
  The POGO score describes the best view of the glottic opening compared to the anatomical picture of the glottis. During direct laryngoscopy the investigator registers an approximate socre, while video laryngoscopy records are assessed by an independent investigator.
Tube insertion time | Registered once during the intubation attempt. Up to 120 seconds following the start of intubation attempt.
  Time necessary for the operator to insert the cuffed endotracheal tube inside the proximal part of the trachea through the glottic opening. Tube insertion time is measured after the investigator finished the search for the glottic opening, achieved best view and decided to insert the tube into the trachea until the cuff is inflated and the airway is secured.
Primary intubation attempt success rate | Measured once after intubation. Up to 120 seconds following the start of intubation attempt.
  All intubation attempts must be finished within 120 seconds or the investigator should give up the attempt and reoxygenize the patient before another attempt. If the investigator finished within the 120 seconds time frame we assess endotracheal tube position by capnography and auscultation. The attempt is regarded successful if the tube is in the right position and the airway is secured.

CONTACTS AND LOCATIONS:
Overall Officials: Bálint Nagy, MD PhD, Study Chair — Department of Anesthesiology and Intensive Therapy, University of Pécs, Hungary; Szilárd Rendeki, MD, Study Chair — Department of Anesthesiology and Intensive Therapy, University of Pécs, Hungary; Lajos Bogár, MD PhD DSc, Study Chair — Department of Anesthesiology and Intensive Therapy, University of Pécs, Hungary
Locations (1):
- University of Pécs, Dept. of Anaesthesia and Intensive Care, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rendeki S, Keresztes D, Woth G, Merei A, Rozanovic M, Rendeki M, Farkas J, Muhl D, Nagy B. Comparison of VividTrac(R), Airtraq(R), King Vision(R), Macintosh Laryngoscope and a Custom-Made Videolaryngoscope for difficult and normal airways in mannequins by novices. BMC Anesthesiol. 2017 May 26;17(1):68. doi: 10.1186/s12871-017-0362-y. PMID 28549421